CLINICAL TRIAL: NCT07245511
Title: A Prospective Observational Study Comparing the VIDIAC, PeDiAC, and Intubation Difficulty Scale (IDS) in Pediatric Patients Aged 5-18 Years Undergoing Tracheal Intubation With Videolaryngoscopy
Brief Title: Comparison of VIDIAC, PeDiAC and Intubation Difficulty Scale in Pediatric Patients Undergoing Videolaryngoscopic Intubation
Acronym: VIDIPEDIDS
Status: Recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: VIDIPEDIIDS-25
Record Dates: First submitted 2025-09-24; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Videolaryngoscopy; Intubation Difficulty Scale; Vidiac Score; Difficult Airway Intubation; Pediatric Anesthesia
Keywords: intubation difficulty scale (IDS); VIDIAC; PeDiAC; Pediatric anesthesia; videolaryngoscopy; airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients Undergoing Videolaryngoscopic Intubation: This cohort will include pediatric patients aged 5 to 18 years undergoing elective or emergency surgery under general anesthesia who require tracheal intubation. All patients will be intubated using a C-MAC videolaryngoscope. Each intubation will be evaluated using the VIDIAC, PeDiAC, and Intubation Difficulty Scale (IDS) scoring systems.

SUMMARY:
This prospective observational study aims to evaluate three scoring systems (VIDIAC (Video Laryngoscopic Intubation and Difficult Airway Classification), PeDiAC (Pediatric Difficult Airway Classification), and the Intubation Difficulty Scale (IDS)).

A total of 450 children undergoing general anesthesia with videolaryngoscopic intubation will be included in the study. Demographic data, intraoperative parameters, and glottic imaging, as well as detailed intubation-related variables such as total intubation time, number of attempts, complications, and subjective intubation ease scores will be recorded.

DETAILED DESCRIPTION:
This study is a prospective, observational, single-center study designed to compare three difficult intubation scales (VIDIAC [Video Laryngoscopic Intubation and Difficult Airway Classification], PeDiAC [Pediatric Difficult Airway Classification], and the Intubation Difficulty Scale [IDS]).

A total of 450 children undergoing elective or emergency surgery under general anesthesia at Ankara Bilkent City Hospital will be included in the study. All tracheal intubations will be performed using a C-MAC videolaryngoscope with an endotracheal tube appropriate for the child's age, weight, and surgical indication. No procedures beyond routine clinical practice will be performed, and informed consent will be obtained from parents or legal guardians prior to inclusion in the study.

Data collection will include demographic characteristics (age, gender, weight, height, ASA classification, comorbidities), intraoperative parameters (SpO₂, heart rate), and intubation-related variables: Glottic view graded using the modified Cormack-Lehane classification, time required for glottic visualization, total intubation time, number of attempts, use of adjuncts (stylet, bougie, alternative tubes), complications (desaturation, esophageal intubation, mucosal bleeding, tooth or lip trauma).

This study will evaluate difficult tracheal intubation in pediatric patients aged 5 to 18 years. Three difficult intubations The difficulty of intubation will be rated subjectively (0 = extremely easy, 10 = impossible) by the anesthesiologist performing the intubation and independently by an observer.

ELIGIBILITY:
Eligible participants will be pediatric patients aged 5 to 18 years who are undergoing general anesthesia for any surgical procedure. All included patients must undergo tracheal intubation using a videolaryngoscope (C-MAC). Patients must have an ASA physical status classification of I to IV and written informed consent must be obtained from a parent or legal guardian prior to participation.

Inclusion Criteria:

* Pediatric patients between 5 and 18 years of age
* Undergoing general anesthesia for any type of surgical procedure
* ASA physical status classification I to IV
* Written informed consent obtained from parents or legal guardians

Exclusion Criteria:

* Patients undergoing awake fiberoptic intubation
* History of tracheal resection or reconstruction surgery
* Refusal to participate or absence of informed consent

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This study will include pediatric patients aged 5 to 18 years who are scheduled for elective or emergency surgery under general anesthesia at Ankara Bilkent City Hospital. All participants will require tracheal intubation performed with a C-MAC videolaryngoscope. Eligible patients will have an ASA physical status classification of I-IV. Written informed consent will be obtained from parents or legal guardians prior to enrollment. Patients undergoing awake fiberoptic intubation, those with a history of tracheal resection, or children younger than 5 years will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Comparison of VIDIAC, PeDiAC, and IDS Scores in the Evaluation of Difficult Intubation in Children | Immediately after tracheal intubation
  For each patient, VIDIAC, PeDiAC, and Intubation Difficulty Scale (IDS) scores will be calculated immediately after tracheal intubation via videolaryngoscopy. These scores will be statistically analyzed to determine the correlation between the number of intubation attempts, intubation time, complications, and subjective intubation ease ratings, in order to identify the scoring system that provides the most reliable assessment of difficult intubation in children.
A Prospective Observational Study Comparing VIDIAC, PeDiAC, and the Intubation Difficulty Scale (IDS) in Assessing Difficult Intubation in Pediatric Patients Aged 5-18 Years Undergoing Tracheal Intubation with Videolaryngoscopy | Immediately after tracheal intubation
  For each patient, VIDIAC, PeDiAC, and Intubation Difficulty Scale (IDS) scores will be calculated immediately after tracheal intubation via videolaryngoscopy. These scores will be statistically analyzed to determine the correlation between the number of intubation attempts, intubation time, complications, and subjective intubation ease ratings, in order to identify the scoring system that provides the most reliable assessment of difficult intubation in children.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Department Of Anesthesiology and Reanimation, Ankara, Turkiye, Turkey (Türkiye)